CLINICAL TRIAL: NCT06149000
Title: Migraine Headache Mitigation Utilizing Avulux Color Filtering Lenses
Brief Title: Migraine Headache Mitigation Utilizing Avulux
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Avulux
Record Dates: First submitted 2023-11-01; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Migraine; Headache; Photophobia
MeSH Terms: conditions — Migraine Disorders; Headache; Photophobia

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, double blind, crossover interventional trial. Participants will be randomly assigned to one of 2 groups of 20. 1. Experimental Group: Participants in this group will wear Avulux lenses during the testing sessions. 2. Control Group: Participants in this group will wear placebo lenses that resemble Avulux lenses but do not have the same optical properties.
Who Masked: Participant, Investigator
Masking Description: Neither the participants or the researchers will know which treatment is being received during the trial. This will be achieved by using identical looking placebos for control and ensuring all aspects of the treatment administration and assessment are indistinguishable.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Avulux Lenses (Experimental): This group will be receiving migraine treatment using Avulux lenses
  Interventions: Device: Avulux Lenses; Device: Placebo Lenses
- Placebo Lenses (Placebo Comparator): This group will be using identical placebo lenses as treatment
  Interventions: Device: Avulux Lenses; Device: Placebo Lenses

INTERVENTIONS:
Device: Avulux Lenses — Avulux lenses are specialized eyewear designed to reduce specific wavelengths of light to alleviate symptoms in individuals who experience light sensitivity and migraines
Device: Placebo Lenses — Lenses that will look identical to Avulux lenses without the medical benefits

SUMMARY:
This will be a randomized double blind cross over interventional trial to determine if Avulux lenses are able to reduce headache symptoms in patients

DETAILED DESCRIPTION:
Participants:

This study will include a total of 40 participants aged 18 and over who have been screened for migraine headache history. Patients who attended the SBC Headache class with a diagnosis of Migraine from the last 12 months will be selected and assigned a number. Random number set will be used to select the 40 patients. Additional 40 patients will be selected to meet the total initial enrollment of 40 patients in the end. These 40 patients will be randomly assigned to Avulux or Control groups. Each patient will be assigned a unique identifier, and the rest of the correspondents will not use patient demographics.

Design:

The study will be a randomized, double blind, crossover interventional trial. Participants will be randomly assigned to one of 2 groups of 20. 1. Experimental Group: Participants in this group will wear Avulux lenses during the testing sessions. 2. Control Group: Participants in this group will wear placebo lenses that resemble Avulux lenses but do not have the same optical properties.

Procedure:

Participants will complete a baseline assessment and self-report migraine frequency using the Redcap migraine diary application. Participants will complete testing sessions with both Avulux and placebo lenses for the duration of 3 months and then switch lenses for the remaining 3 months for comparison and a total study period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient population: Individuals must have an existing diagnosis code of G43.1 (migraine w aura) or G43. 10 (migraine w aura, not intractable).
* Only Kaiser Permanente members receiving care at the Fontana Medical Service Areas will be in consideration.
* Patients that are >18
* There will no restrictions based on biological sex.
* Participants will be referred to optical by provider (Neurologists/Optometrist/Primary Care physician).
* Participants must agree to not initiate any new medical management during the trial or be willing to voluntarily withdrawal from participating in the trial

Exclusion Criteria:

* Patients who do not have a migraine diagnosis code in their medical record.
* Patients that have started a new migraine medication within last 30 days
* Non-Members of Kaiser Permanente

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-13 (Estimated); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Reduction in migraine frequency | 6 months
  headache days per month documented in a headache diary.
Reduction in migraine severity | 6 months
  Severity of headaches on a scale from no, mild, moderate, and sever pain

SECONDARY OUTCOMES:
Improve quality of life | 6 months
  Rating of daily activity performance using Functional Disability Scale (0) No disability-(6) Severe disability
Medication Use | 6 months
  Number of medications used as a form of rescue medication during episode of migraine

CONTACTS AND LOCATIONS:
Overall Officials: Munish Sharma, OD/MBA, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared

REFERENCES:
- [Background] Posternack C, Kupchak P, Capriolo AI, Katz BJ. Targeting the intrinsically photosensitive retinal ganglion cell to reduce headache pain and light sensitivity in migraine: A randomized double-blind trial. J Clin Neurosci. 2023 Jul;113:22-31. doi: 10.1016/j.jocn.2023.04.015. Epub 2023 May 5. PMID 37150129
- [Background] Katz BJ, Digre KB. Diagnosis, pathophysiology, and treatment of photophobia. Surv Ophthalmol. 2016 Jul-Aug;61(4):466-77. doi: 10.1016/j.survophthal.2016.02.001. Epub 2016 Feb 12. PMID 26875996
- [Background] Wilkins AJ, Wilkinson P. A tint to reduce eye-strain from fluorescent lighting? Preliminary observations. Ophthalmic Physiol Opt. 1991 Apr;11(2):172-5. doi: 10.1111/j.1475-1313.1991.tb00217.x. PMID 2062542
- [Background] Huang J, Zong X, Wilkins A, Jenkins B, Bozoki A, Cao Y. fMRI evidence that precision ophthalmic tints reduce cortical hyperactivation in migraine. Cephalalgia. 2011 Jun;31(8):925-36. doi: 10.1177/0333102411409076. Epub 2011 May 26. PMID 21622479
- See also: Avulux Migraine and Light Sensitivity Pilot Study Published in the Journal of Clinical Neuroscience — https://pubmed.ncbi.nlm.nih.gov/26935748/
- See also: Avulux Randomized Trial — https://clinicaltrials.gov/ct2/show/NCT04341298